CLINICAL TRIAL: NCT07196956
Title: The Role of Electromagnetic Field Therapy in Improving Perturbation of Balance and Gait Disorders in Paraparetic Patients
Brief Title: Effect of Electromagnetic Field Therapy on Balance and Gait in Paraparetic Patients
Acronym: EMT-BG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, reda abd elrazik, Associate Professor, Department of Physical Therapy for musculoskeletal disorders and its surgery, Faculty of Physical Therapy, Benha University, MTI University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT. BU. EC. 28
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Paraparesis; Gait Disorders, Neurologic; Postural Balance Disorders
Keywords: Electromagnetic Field Therapy; Electromagnetic Stimulation; Physical Therapy Modalities; Spasticity; Rehabilitation; Biodex Balance System; Motion Analysis; Modified Ashworth Scale
MeSH Terms: conditions — Paraparesis; Gait Disorders, Neurologic; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Thirty paraparetic patients will be randomly assigned to one of two parallel groups. Group I will receive a placebo electromagnetic therapy device plus a standard physical therapy program. Group II will receive active electromagnetic field therapy plus the identical physical therapy program.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the active and placebo electromagnetic therapy devices will appear identical to participants and study personnel. The settings on the devices will be controlled by an independent technician not involved in patient care or outcome assessment to ensure blinding of participants, care providers, investigators, and outcomes assessors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo EMT + Physical Therapy (Placebo Comparator): Participants will receive a placebo (inactive) electromagnetic therapy device applied to the spine, combined with a standardized 45-minute physical therapy program. The physical therapy program includes stretching exercises, strengthening exercises, balance training, and gait training. Treatment will be administered three times per week for 2 months.
  Interventions: Device: Placebo Electromagnetic Field Therapy
- Active EMT + Physical Therapy (Experimental): ticipants will receive active low-frequency (0.5 Hz) electromagnetic field therapy applied to the spine, combined with the identical 45-minute physical therapy program (stretching, strengthening, balance, and gait training) as the control group. Treatment will be administered three times per week for 2 months.
  Interventions: Device: Low-Frequency Electromagnetic Field Therapy (0.5 Hz)

INTERVENTIONS:
Device: Low-Frequency Electromagnetic Field Therapy (0.5 Hz) — Active electromagnetic field therapy delivered via a PMT Quattro PRO device (Italy, 2002). Settings: 0.5 Hz frequency, 30 mA intensity, applied for 20 minutes per session to the spinal lesion level (T6-T12) while patient is prone. Followed by 10-minute rest. Administered three times per week for 2 months, in conjunction with a standardized 45-minute physical therapy program (stretching, strengthening, balance, and gait training).
  Other Names: EMT,; Pulsed Electromagnetic Field Therapy
  Arms: Active EMT + Physical Therapy
Device: Placebo Electromagnetic Field Therapy — identical-appearing electromagnetic therapy device with no active field output (placebo/sham). Applied for 20 minutes per session to the spinal lesion level (T6-T12) while patient is prone. Followed by 10-minute rest. Administered three times per week for 2 months, in conjunction with the identical standardized 45-minute physical therapy program (stretching, strengthening, balance, and gait training) as the active EMT group.
  Other Names: Sham EMT; Inactive EMT
  Arms: Placebo EMT + Physical Therapy

SUMMARY:
This study will investigate whether adding electromagnetic field therapy (EMT) to a standard physical therapy program is more effective than physical therapy alone for improving balance and walking ability in paraparetic patients.

Thirty patients with paraparesis (weakness in the lower limbs) due to spinal cord lesions between levels T6 and T12 will be randomly assigned to one of two groups. Both groups will receive a 45-minute physical therapy session, three times per week for two months. The physical therapy program will include stretching, strengthening, balance, and gait training exercises.

The key difference will be that one group (Group II) will also receive active low-frequency (0.5 Hz) electromagnetic therapy applied to their spine during their sessions, while the other group (Group I) will receive a placebo (inactive) EMT device.

Patients will be assessed before and after the 2-month treatment period. The assessments will measure muscle spasticity (using the Modified Ashworth Scale), balance (using the Biodex Balance System), and detailed gait parameters like step length, stride length, and base of support (using a 3D motion analysis system

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of paraparesis with spinal cord lesion level between T6 and T12. Age between 25 and 45 years. Muscle spasticity graded as II or III on the Modified Ashworth Scale (MAS) for hip adductors and ankle plantar flexors.

Medically and psychologically stable. Conscious and cooperative, able to follow instructions. Able to provide informed consent.

Exclusion Criteria:

* Presence of metal implants or pacemakers (contraindicated for electromagnetic therapy).

History of seizures or epilepsy. Active malignancy or infection. Severe cognitive or psychiatric impairment that would interfere with participation.

Use of alcohol or recreational drugs during the study period. Participation in another concurrent physical or electromagnetic therapy trial. Unstable medical condition (e.g., uncontrolled hypertension, cardiovascular disease).

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-11 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Spasticity as Measured by the Modified Ashworth Scale (MAS) | Baseline (pre-treatment) and at 2 months (post-treatment)
  Spasticity of the hip adductor and ankle plantar flexor muscles will be assessed using the Modified Ashworth Scale (MAS), a 6-point ordinal scale (0 = no increase in muscle tone to 4 = rigid in flexion or extension). The primary comparison will be the change in MAS score from baseline to 2 months between the active EMT group and the placebo EMT group.

SECONDARY OUTCOMES:
Change in Dynamic Balance as Measured by the Biodex Balance System (BBS) | Baseline (pre-treatment) and at 2 months (post-treatment)
  Dynamic postural stability will be assessed using the Biodex Balance System. Participants will perform a single-leg stance test (on the non-dominant leg, eyes closed, hands on hips). The system provides a numerical stability index; a lower score indicates better balance. Change from baseline to 2 months will be compared between groups.
Change in Step Length as Measured by 3D Motion Analysis (Qualisys System) | Step length (distance from heel strike of one foot to heel strike of the opposite foot) will be measured during self-paced walking using the Qualisys 3D Motion Analysis System. The average of three trials will be recorded. Change from baseline to 2 month
  Step length (distance from heel strike of one foot to heel strike of the opposite foot) will be measured during self-paced walking using the Qualisys 3D Motion Analysis System. The average of three trials will be recorded. Change from baseline to 2 months will be compared between groups
Change in Stride Length as Measured by 3D Motion Analysis (Qualisys System) | Baseline (pre-treatment) and at 2 months (post-treatment)
  Stride length (distance from heel strike of one foot to the next heel strike of the same foot) will be measured during self-paced walking using the Qualisys 3D Motion Analysis System. The average of three trials will be recorded. Change from baseline to 2 months will be compared between groups.
Change in Base of Support as Measured by 3D Motion Analysis (Qualisys System) | Baseline (pre-treatment) and at 2 months (post-treatment)
  Base of support (lateral distance between the left and right feet during walking) will be measured during self-paced walking using the Qualisys 3D Motion Analysis System. The average of three trials will be recorded. Change from baseline to 2 months will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic, Department of Physical Therapy, Faculty of Applied Medical Science, Najran University, Najrān, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided